CLINICAL TRIAL: NCT01658267
Title: Compliance With Dietary Recommendations in Meeting Nutritional Requirements in Children at Risk of Undernutrition
Brief Title: Compliance With Dietary Recommendations in Children at Risk for Undernutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK86
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Children; Under-nutrition
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional Supplement (Experimental): Instructions and techniques to improve the quality of the diet to meet the child's daily nutritional requirements will be provided.
  Interventions: Other: nutritional supplement

INTERVENTIONS:
Other: nutritional supplement — 2 servings per day
  Other Names: Pediasure S229

SUMMARY:
This study will assess compliance with dietary recommendations, in conjunction with a nutritional supplement to meet the nutritional requirements in children and the effects of the compliance on promoting growth in children who are at risk of under-nutrition.

DETAILED DESCRIPTION:
This study will assess compliance with dietary recommendations, in conjunction with an oral nutritional supplement to meet the nutritional requirements in children older than 36 (>36) to less than or equal 48 (≤48) months of age, and the effects of the compliance on promoting catch-up growth and normal healthy growth in children who are at risk of under-nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 36 and 48 months of age.
* Child has weight-for-height greater than or equal to 5th and less than or equal to the 25th percentile.
* Child is capable of oral feeding.
* Child's parent(s)or Legal Guardian is willing to abstain from giving additional non-study nutritional supplements to the child throughout the study period.

Exclusion Criteria:

* Child whose either parent has BMI greater than or equal to 27.5 kg/m2.
* Child allergic or intolerant to any ingredient found in the study product.
* Child who was delivered pre-term.
* Child was born small for gestational
* Child had birth weight < 2500 g or > 4000 g.
* Child has current acute or chronic infections.
* Child demonstrates presence of severe gastrointestinal disorders.
* Child has a diagnosis of neoplastic diseases, renal, hepatic and cardiovascular diseases.
* Child has a diagnosis of hormonal or metabolic disorders.
* Child has a congenital disease or genetic disorder.
* Child is diagnosed with infantile anorexia nervosa.
* Child has a developmental disability or physical disorder.
* Child has disorders of hemoglobin structure, function or synthesis.
* Child is participating in another study that has not been approved as a concomitant study.

Ages: 36 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Compliance with recommendation of a nutritional supplement consumption | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dieu Huynh, MD, PhD, Study Chair — Abbott Nutrition, Singapore
Locations (2):
- Philippines (2):
  - Asian Hospital and Medical Center, Manila
  - The Medical City, Manila